CLINICAL TRIAL: NCT04550247
Title: A National, Prospective, Non- Interventional Study (NIS) in Patients Receiving Adjuvant Nivolumab Therapy for Resected Melanoma and Subsequent Treatments in Case of Relapse
Brief Title: A Prospective Non-Interventional Study in Participants Receiving Nivolumab in Adjuvant Setting for Resected Melanoma in Real-World Conditions in France
Acronym: AdjuMel
Status: Active, not recruiting | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: CA209-7HU
Record Dates: First submitted 2020-09-09; First posted 2020-09-16 (Actual); Last update posted 2022-03-21 (Actual); Status verified 2022-03

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Nivolumab treatment: Administered according to the market authorization in France

SUMMARY:
This is an observational prospective study to estimate in real world conditions the effectiveness, the safety profile and the pattern of use of adjuvant nivolumab in adults participants with stage III/IV resected melanoma, and subsequent treatments administered in case of relapse.

ELIGIBILITY:
For more information regarding Bristol-Myers Squibb Clinical Trial participation,please visit www.BMSStudyConnect.com.

Inclusion Criteria:

* Participants with a primary diagnosis of melanoma with involvement of lymph nodes or metastatic disease who have undergone complete resection and have no evidence of disease
* Decision to treat with adjuvant nivolumab therapy has already been taken
* Participants who provide oral informed consent to participate in the study

Exclusion Criteria:

* Any participant with a current diagnosis of persisting advanced melanoma
* Participants with a current primary diagnosis of a cancer other than advanced melanoma, ie, a cancer other than melanoma that requires systemic or other treatment or has not been treated curatively (as per discretion of the investigator)
* Any participants currently enrolled in an interventional clinical trial for his/her melanoma treatment (note: patients who have completed their participation in an interventional trial or who are no longer receiving the study drug and are only followed up for OS/RFS can be enrolled. In case of a blinded study, the treatment arm needs to be known).
* Pregnant women
* Person under guardianship

Other protocol defined inclusion/exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will collect data primarily from hospital based dermatology and oncology care facilities
Sampling Method: Non-Probability Sample
Enrollment: 362 (Actual)
Dates: Start 2020-09-02 (Actual); Primary Completion 2027-03-15 (Estimated); Study Completion 2027-03-15 (Estimated)

PRIMARY OUTCOMES:
Relapse-Free Survival (RFS) | up to 60 months

SECONDARY OUTCOMES:
Distant Metastatasis-Free Survival (DMFS) | Up to 60 months
Overall Survival (OS) | Up to 60 months
Relapse-Free Survival 2 (RFS2) | Up to 60 months
Progression Free Survival (PFS) | Up to 60 months
Assessment of health related quality of life | Up to 60 Months
Assessment of sociodemographic characteristics | Up to 60 months
Assessment of clinical characteristics | Up to 60 months
Frequency of nivolumab therapy: number of infusions | Up to 60 months
Frequency of nivolumab therapy: number of dosing | Up to 60 months
Frequency of Nivolumab: pattern of use | Up to 60 months
Characteristics of nivolumab adjuvant safety profile: incidence | Up to 60 months
Characteristics of nivolumab adjuvant safety profile: grade | Up to 60 months
Characteristics of nivolumab adjuvant safety profile: type | Up to 60 months
Characteristics of nivolumab adjuvant safety profile: time to onset of select AEs | Up to 60 months
Characteristics of nivolumab adjuvant safety profile: time to onset of other immune- related AEs | Up to 60 months
Characteristics of nivolumab adjuvant safety profile: time to resolution of select AEs | Up to 60 months
Characteristics of nivolumab adjuvant safety profile: time to resolution of other immune-related AEs | Up to 60 months
Describe the use of subsequent therapies after relapse following adjuvant nivolumab | Up to 60 months
Estimate of the effectiveness of systemic therapies administered after relapse following adjuvant nivolumab, in terms of time and duration of response | Up to 60 months
Estimate of the effectiveness of systemic therapies administered after relapse following adjuvant nivolumab, in terms of overall response rate | Up to 60 months
Safety profile of systemic therapies administered after relapse in terms of severe adverse events incidence, type, management and outcome | Up to 60 months
Estimate the effectiveness of subsequents treatments administered after relapse in terms of PFS | Up to 60 months
Estimate the effectiveness of subsequents treatments administered after relapse in terms of RFS2 | Up to 60 months
Estimate the effectiveness of subsequents treatments administered after relapse in terms of OS | Up to 60 months
Characteristics of nivolumab adjuvant safety profile: management | Up to 60 months
Characteristics of nivolumab adjuvant safety profile: outcome | Up to 60 months
Safety profile of systemic therapies administered after relapse in terms of severe adverse events: Incidence | Up to 60 months
Safety profile of systemic therapies administered after relapse in terms of severe adverse events: Type | Up to 60 months
Safety profile of systemic therapies administered after relapse in terms of severe adverse events: Management | Up to 60 months
Safety profile of systemic therapies administered after relapse in terms of severe adverse events: Outcome | Up to 60 months

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution, Lille, France

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/investigator-inquiry-form.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm